CLINICAL TRIAL: NCT07166666
Title: Study Comparing Atomizerd Midazolam & Fentanyl and Dexmedomidine for Procedural Sedation in Adult and Pediatric Patient (2 to 60 Years Old)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Ghaliya Al Noofli, Principal Investigator, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MoH/CSR/24/28497; MOH/ oman (Other: MOH)
Record Dates: First submitted 2025-07-23; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Sedation; Analgesia Assessment
MeSH Terms: interventions — Nebulizers and Vaporizers; Midazolam; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- midazolame $ fentanyl (Other): use as compare between two group
  Interventions: Device: atomizer; Drug: rescue medication; Drug: Midazolam; Drug: fentanyl
- dexetomidate (Other): use as compare to other group
  Interventions: Device: atomizer; Drug: rescue medication; Drug: Dexmedetomidine; Drug: Placabo

INTERVENTIONS:
Device: atomizer — use atomizer to provide the medication in procedure sedation
Drug: rescue medication — will be used as rescue if the atomizer medication not fully sedated
Drug: Midazolam — Intranasal administration for procedural sedation.
  Arms: midazolame $ fentanyl
Drug: fentanyl — Intranasal administration for procedural sedation.
  Arms: midazolame $ fentanyl
Drug: Dexmedetomidine — Intranasal administration for procedural sedation.
  Arms: dexetomidate
Drug: Placabo — use atomizer to provide the placebo in procedure sedation
  Arms: dexetomidate

SUMMARY:
To evaluate the depth of sedation, as well as onset, and recovery times, satisfaction of sedation , adverse events associated with Atomized Midazolam & Fentanyl and Dexmedetomidine during procedural sedation in a diverse population spanning from 2 to 60 years old at these three prominent Omani healthcare facilities.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria:

  1. Patients aged 2 to 60 years.
  2. Patients undergoing EM procedures requiring sedation.

Exclusion criteria:

1. Patients with contraindications to any of the sedation agents being studied.
2. Patients with a history of adverse reactions or allergies to the study medications.
3. Drug interactions: Patients taking certain medications that may interact adversely with the study medications.
4. Drug Abuser
5. Pregnancy and breastfeeding
6. Patients with significant cardiovascular or respiratory compromise.
7. Patients with nasal disorder (nasal trauma, epistaxis)
8. Patients unable to provide informed consent or those with cognitive impairment.
9. Patients who are < 2 year of age or > 60 year of age.
10. Patient underwent procedure sedation for imaging

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
depth of sedtion | 1 year
  using MOAA/S score, Modified Observer's Assessment of Alertness/Sedation Scale , as 0 high score for deep sedation, 5 not in deep sedation

CONTACTS AND LOCATIONS:
Overall Officials: saud al bulashi, MD, Study Director — MOH/ oman
Locations (1):
- dr.Suad al baluish, Muscat, Oman